CLINICAL TRIAL: NCT03101046
Title: Personalized Treatment of Metastatic Castrate Resistant Prostate Cancer Patients According to Circulating Tumor Cells Kinetic During Chemotherapy: A GETUG-AFU 28 Study
Brief Title: Treatment of Metastatic Castrate Resistant Prostate Cancer Patients According to Circulating Tumor Cells Kinetic
Acronym: TACTIK
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UNICANCER (Other)
Collaborators: National Cancer Institute, France (Other Government); Institut du Cancer de Montpellier - Val d'Aurelle (Other); Institut Bergonié (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GETUG-AFU-28 - UC-0160/1613; 2016-002429-12 (EudraCT Number)
Record Dates: First submitted 2017-03-22; First posted 2017-04-04 (Actual); Last update posted 2022-02-10 (Actual); Status verified 2022-02

CONDITIONS: Prostate Carcinoma; Castration-resistant Prostate Cancer; Circulating Tumor Cells; Chemotherapy
Keywords: Docetaxel; Cabazitaxel
MeSH Terms: conditions — Prostatic Neoplasms; Neoplastic Cells, Circulating | interventions — cabazitaxel; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group1: Arm A (standard arm) + Arm B (experimental arm) (Other): Arm A: Patients with docetaxel resistant mCRPC (defined as having ≥5 CTCs / 7.5 mL) will receive up to 8 additional cycles of docetaxel (75 mg/m² every 3 weeks) after randomization.
  Arm B: Patients with docetaxel resistant mCRPC (defined as having ≥5 CTCs / 7.5 mL) will receive up to 10 cycles of cabazitaxel (20 mg/m² every 3 weeks) after randomization.
  Interventions: Drug: Cabazitaxel; Drug: Docetaxel
- Group 2: Cohort (Other): Patients with docetaxel sensitive mCRPC (defined as having <5 CTCs / 7.5 mL) will receive up to 8 additional cycles of docetaxel (75 mg/m² every 3 weeks)
  Interventions: Drug: Docetaxel

INTERVENTIONS:
Drug: Cabazitaxel — Experimental treatment arm: patients will be treated with intravenous cabazitaxel 20 mg/m² every 3 weeks up to 10 cycles.
  Other Names: JEVTANA
  Arms: Group1: Arm A (standard arm) + Arm B (experimental arm)
Drug: Docetaxel — standard treatment arm and cohort: Docetaxel is administered at the dose of 75 mg/m² over 1 hour every 3 weeks for 6 cycles (D1=D22).

SUMMARY:
This study compares the biological activity of cabazitaxel (6 cycles) to that of docetaxel (6 cycles) in metastatic castrate-resistant prostate cancer (mCRPC) patients with docetaxel resistant mCRPC defined as ≥5 circulating tumor cells (CTCs) / 7.5 mL after 2 cycles of docetaxel.

Patients with docetaxel resistant metastatic castration-resistant prostate cancer (mCRPC) based on circulating tumor cell (CTC) enumeration (patients with ≥5 CTCs / 7.5 mL before docetaxel chemotherapy and after 2 cycles of docetaxel) will receive either 6 additional cycles of docetaxel or 6 additional cycles of cabazitaxel after randomisation.

A cohort of patients with docetaxel sensitive metastatic castration-resistant prostate cancer (mCRPC) based on circulating tumor cell (CTC) enumeration (patients ≥5 CTCs / 7.5 mL before docetaxel chemotherapy and <5 CTCs / 7.5 mL after 2 cycles of docetaxel) will receive 6 additional cycles of docetaxel.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent signed prior any study-related procedures
2. Adult men ≥18 years
3. Histologically confirmed prostate adenocarcinoma
4. Metastatic disease as evidenced by imaging (bone scan, CT-scan, MRI and/or PET-choline).
5. Documented progressive disease while receiving continuous hormonal treatment with luteinizing hormone-releasing hormone (LH-RH) agonist or antagonist or after surgical castration (at least one visceral or soft tissue metastatic lesion, including a new lesion). Patient with non-measurable disease must have documented rising prostate-specific antigen (PSA) levels or appearance of new lesion
6. Effective castration assessed by testosterone levels ≤50 ng/dL
7. Patients with a Eastern Cooperative Oncology Group (ECOG) performance status ≤2
8. Patients affiliated to social security scheme

Exclusion Criteria:

1. Prior chemotherapy for metastatic prostate cancer except estramustine <1 year from the end of adjuvant and/or neoadjuvant chemotherapy for localized disease <1 year from the end of chemotherapy for de novo metastatic prostate cancer
2. Prior isotope therapy, whole pelvic radiotherapy or radiotherapy to >30% of bone marrow
3. Less than 1 month elapsed from prior treatment with radiotherapy, surgery and less than 2 weeks from any previous hormonal treatment except for LH-RH agonists/antagonists (which are to be continued). Patients may be treated with bisphosphonates prior to study entry which should be pursued,
4. History of brain metastases, uncontrolled spinal cord compression, carcinomatous meningitis or new evidence of brain or leptomeningeal disease
5. Patient with any of the following abnormal laboratory tests: hemoglobin <10 g/dL, absolute neutrophil count <1.5 x 10⁹/L, platelets <100 x 10⁹/L, aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) >1.5 x upper limit of normal (ULN), total bilirubin >1.0 ULN, creatinine clearance <40 ml/mn (MDRD)
6. History of hypersensitivity to polysorbate 80 or docetaxel
7. Contraindication to the use of corticosteroids
8. Peripheral neuropathy grade ≥2 according to NCI CTCAE v4.0
9. Ventricular ejection fraction <50% (echography or scintigraphy)
10. Any of the following within 6 months prior to study entry: myocardial infarction, severe/unstable angina pectoris, coronary/peripheral artery bypass graft, New York Heart Association (NYHA) class III or IV congestive heart failure, stroke or transient ischemic attack
11. Any of the following within 3 months prior to study entry: treatment resistant peptic ulcer disease, erosive esophagitis or gastritis, inflammatory bowel disease, pulmonary embolism or other uncontrolled thromboembolic event
12. Other severe acute or chronic medical or psychiatric condition, or laboratory abnormally that would impart, in the judgment of the investigator, excess risk associated with study participation or study drug administration, or which, in the judgment of the investigator, would make the patient inappropriate for entry into this study
13. Planned vaccination with a live or live-attenuated vaccines
14. Participation in another clinical trial and any treatment with any investigational drug within 30 days prior to randomization
15. Any illness or problem including geographic, psychiatric or psychological which is incompatible with being monitored during the trial
16. Patients with reproductive potential who do not agree to use effective method of contraception during the treatment
17. Person deprived of their liberty or under protective custody or guardianship

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-11-15 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Biological activity of chemotherapy | 18 weeks after randomisation
  Biological activity of chemotherapy as defined as < 5 CTCs per 7.5 ml at the end of chemotherapy with docetaxel or cabazitaxel.

CONTACTS AND LOCATIONS:
Overall Officials: Stéphane CULINE, Principal Investigator — Hôpital Saint Louis Paris
Locations (5):
- France (5):
  - ICO-Site Paul Papin, Angers
  - CHD Vendée, La Roche-sur-Yon
  - Centre Léon Berard, Lyon
  - Stéphane CULINE, Paris
  - ICO-Site René Gauducheau, Saint-Herblain

IPD SHARING:
Plan to Share IPD: No